CLINICAL TRIAL: NCT04683718
Title: BENEFIT-03 Clinical Study
Brief Title: A First in Human Feasibility Study to Evaluate the Safety and Effectiveness of the BIOTRONIK Prospera SCS System with HomeStream Remote Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Collaborators: Biotronik Australia Pty Ltd. (Industry); BIOTRONIK Neuro (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BENEFIT-03
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Chronic Low-back Pain; Chronic Leg Pain
MeSH Terms: interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BIOTRONIK Prosper SCS (Spinal Cord Stimulation) System (Experimental): Eligible participants will be permanently implanted with a BIOTRONIK Prospera SCS (Spinal Cord Stimulation) System with HomeStream Remote Management.
  Interventions: Device: Permanent implant of a BIOTRONIK Prospera SCS (Spinal Cord Stimulation) System with HomeStream Remote Management

INTERVENTIONS:
Device: Permanent implant of a BIOTRONIK Prospera SCS (Spinal Cord Stimulation) System with HomeStream Remote Management — The Prospera SCS System is a rechargeable, 16-electrode, MRI conditional Spinal Cord Stimulation system that delivers electrical stimulation to the dorsal column of the spinal cord for the treatment of chronic intractable pain of the trunk and/or limbs.

SUMMARY:
The BENEFIT-03 Clinical Study is a first in human, prospective, multi-center, single-arm, interventional feasibility study to be conducted in Australia. The purpose of the BENEFIT-03 study is to collect initial safety and effectiveness data on the BIOTRONIK Prosper SCS (Spinal Cord Stimulation) System with HomeStream Remote Management. Enrolled participants will complete a SCS trial period per the standard of care utilizing the BIOTRONIK Resilience percutaneous SCS trial leads and the BIOTRONIK Prospera External Pulse Generator (EPG). Following a successful trial period, participants will be implanted with a permanent BIOTRONIK Prospera Implantable Pulse Generator (IPG). Implanted participants will be followed for 24 months post-implant with in-office visits and remote management visits.

ELIGIBILITY:
Inclusion Criteria:

* Currently indicated for SCS therapy for the treatment of low back and/or leg pain
* Planned permanent implant of BIOTRONIK's Prospera SCS System with HomeStream Remote Management
* Planned placement of two BIOTRONIK Resilience SCS trial leads
* Documented scores of ≥ 60 mm out of 100 mm on the Visual Analog Scale (VAS) for both overall pain intensity and pain intensity in the index area of pain, assessed at the time of enrollment
* Willing and able to comply with all study requirements, including all required procedures, phone and/or video calls, and study visits
* Age greater than or equal to 18 years and less than 80 years
* Able to understand the nature of the study and provide written informed consent
* Able to read, understand, and speak English
* Patient's pain-related medication regimen is stable 4 weeks prior to the baseline evaluation
* Oswestry Disability Index (ODI) score of 41 to 80 out of 100
* Passed psychological evaluation
* For diabetic patients: minimum of one HbA1c test within the last 6 months, with most recent result ≤ 8.0%

Exclusion Criteria:

* Any contraindication for SCS therapy
* Patients with an implanted pacemaker, defibrillator, or any other medical contraindication for SCS therapy
* Currently implanted with an infusion pump or any implantable neurostimulator device
* Previously implanted with a neurostimulation system or prior participation in a trial period for a neurostimulation system
* Currently enrolled in any investigational device or drug trial for the management of chronic pain
* Patients who have undergone spinal surgery within 12 months prior to enrollment
* Patients currently involved in an active WorkCover insurance claim and/or active litigation related to injury associated with indication for SCS
* Patients with a documented history of substance abuse (narcotics, alcohol, etc.) or substance dependency (other than prescribed) in the 6 months prior to enrollment
* Patients currently displaying opioid-seeking behavior
* Presence of any life-threatening, underlying illness
* Life expectancy less than 1 year
* Patients reporting pregnancy at the time of enrollment or intending to become pregnant during the 2-year study duration
* Patients with opioid dosages > 120 morphine milligram equivalents (MME) per day
* Patients with poor compliance for pain management regimen
* Patients with a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the investigator
* Patients with pain originating from peripheral vascular disease
* Current diagnosis of a coagulation disorder or bleeding diathesis
* Patients with a diagnosis of severe thoracic scoliosis that is likely to preclude SCS lead placement
* Patients who are immunocompromised and/or at high risk for infection
* Patients with a documented history of allergic response or sensitivity to material(s) required for the study (e.g. adhesives, titanium, silicone, etc.)

At the conclusion of the trial period, the absence of the following exclusion criteria should be confirmed before proceeding with the permanent Prospera SCS System implant:

* Reduction in overall pain of less than 50% from baseline, assessed using VAS
* Unsuccessful trial period as otherwise determined by the investigator
* Determined by the investigator to be a poor candidate for permanent Prospera SCS System implant per standard of care (e.g. due to infection, non-compliance with pain medication regimen, paresis, clumsiness, numbness, and other)

Additionally, pre-operative screening for staphylococcus aureus (MRSA/MSSA) must be conducted after the SCS trial period and prior to implantation of the permanent device.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Overall Responder Rate to the BIOTRONIK Prospera SCS System Therapy | 6 months post-implant
  The purpose of primary endpoint 1 is to evaluate the overall responder rate of participants to the BIOTRONIK SCS Therapy at the 6-month follow-up interval. To be classified as a responder, a participant must achieve a reduction in overall pain intensity of at least a 50% from baseline, assessed using the Visual Analog Scale (VAS).
Primary Safety Information on the BIOTRONIK Prospera SCS System | 6 months post-implant
  The purpose of primary endpoint 2 is to collect primary safety information on the BIOTRONIK Prospera SCS System from permanent implant through the 6-month follow-up interval.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Verrills, MD, Study Chair — Metro Pain Group
Locations (5):
- Australia (5):
  - Genesis Research Services, Broadmeadow, New South Wales
  - Australian Medical Research, Hurstville, New South Wales
  - Sydney Pain Research Centre, Wahroonga, New South Wales
  - Sunshine Coast Clinical Research, Noosa, Queensland
  - Monash Clinical Research, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: No